CLINICAL TRIAL: NCT05138367
Title: Clinical Study of Human Umbilical Artery Derived Perivascular Stem Cells in the Treatment of Premature Ovarian Failure
Brief Title: Effects of UCA-PSCs in Women With POF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Li-jun Ding (Other)
Responsible Party: Sponsor-Investigator, Li-jun Ding, principal investigator, Nanjing University
Organization: Nanjing University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SZ-POF-2018-12
Record Dates: First submitted 2021-10-28; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Premature Ovarian Failure
Keywords: POF
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UCA-PSC (Experimental): Subsequent to isolation and culture of UCA-PSCs, UCA-PSCs (GMP grade, from Clinical Center for Stem Cell Research of the Affiliated Drum Tower Hospital of Nanjing University Medical School, licensed by the National Institute for China Food and Drug Control) were injected into the ovaries of patients with hormone replacement treatment, which consisted of Premarin (0.625 mg/days on days 1 through 25) combined with Provera (10 mg/day for 10 days a month with monthly withdrawal bleeding).
  Interventions: Procedure: transplantation of human UCA-PSCs or WJ-MSCs into ovaries of POF patients
- WJ-MSC (Experimental): Subsequent to isolation and culture of WJ-MSCs, WJ-MSCs (GMP grade, from Clinical Center for Stem Cell Research of the Affiliated Drum Tower Hospital of Nanjing University Medical School, licensed by the National Institute for China Food and Drug Control) were injected into the ovaries of patients with hormone replacement treatment, which consisted of Premarin (0.625 mg/days on days 1 through 25) combined with Provera (10 mg/day for 10 days a month with monthly withdrawal bleeding).
  Interventions: Procedure: transplantation of human UCA-PSCs or WJ-MSCs into ovaries of POF patients

INTERVENTIONS:
Procedure: transplantation of human UCA-PSCs or WJ-MSCs into ovaries of POF patients — After vaginal sterilization, TVUS-guided transplantation was performed by the senior-level medical physician B Wang), using a SIEMENS ACUSON ANTANES premium edition system (SIEMENS AG Healthcae Sector, Erlangen, Germany), equipped with a 6-10 MHz probe. The solution (a total number of 2×10^7cells, 1×10^7 /400 μL for unilateral ovarian injection) was injected into the ovary by using 21G PTC needles (Hakko Medical Co, Japan) under TVUS guiance. Each patent received up to three transplantations.

SUMMARY:
This study was a single-center randomized controlled trial at the Affiliated Drum Tower Hospital of Nanjing University Medical School. There were patients who underwent clinical follow-ups since 2018 in POF clinic. Patients were given treatment of either UCA-PSC or WJ-MSC.

DETAILED DESCRIPTION:
At entry, all patients had already received a standard non-physiologic hormone replacement regimen. According to blinded preferences for participation, patients were randomized into two treatment groups after an initial 2-month washout period of no therapy. One group received UCA-PSC transplantation plus horone replacement treatment (HRT) (UCA-PSC group), while the other group received WJ-MSC transplantation plus HRT (collagen/WJ-MSC group)

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Premature Ovarian Failure
2. Patients show no response to drug treatment
3. Willing to receive follow up
4. Willing to conceive a baby
5. Age between 18 to 39

Exclusion Criteria:

1. Patients with chromosome abnormalities
2. Patients with congenital ovarian malformations
3. Patients with severe endometriosis
4. Patients with thyroid dysfunction
5. Patients with pregnancy contraindications
6. Patients with hormone replacement therapy contraindications
7. Past history of ovarian tumors or after radiotherapy
8. Can not take the follow-up, or want to take other treatment during the follow-up period
9. Patients with immune system diseases

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Study of POF is only for people whose physical sex is female.
Enrollment: 20 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
blood perfusion in the ovary | within the first 30 weeks (plus or minus 10 weeks) after surgery
  Systolic/Diastolic blood pressure (S/D) value was monitored in bilateral ovaries by transvaginal color Doppler ultrasound detector.
Antral Follicle Diameter | within the first 30 weeks (plus or minus 10 weeks) after surgery
  An antral follicle (or Graafian follicle) is an ovarian follicle during a certain latter stage of folliculogenesis. The antral follicle diameter in the ovaries were record using transvaginal ultrasound scan.

SECONDARY OUTCOMES:
blood flow index in the ovaries | within the first 30 weeks (plus or minus 10 weeks) after surgery
  The blood flow spectrum in bilateral ovaries was monitored by transvaginal color Doppler ultrasound detector, including pulsatility index (PI), resistance index (RI).

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medicine Center, The affiliated Drum Towel Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China